CLINICAL TRIAL: NCT06959225
Title: A Phase 3, Double-Blind, Randomized, Vehicle-Controlled, Efficacy and Safety Study of Ruxolitinib Cream in Participants With Hidradenitis Suppurativa
Brief Title: Study to Evaluate the Efficacy and Safety of Ruxolitinib Cream in Participants With Hidradenitis Suppurativa (TRuE-HS1)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INCB018424-324; 2024-517632-22-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis suppurativa; skin disease; ruxolitinb cream
MeSH Terms: conditions — Hidradenitis Suppurativa; Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ruxolitinib 1.5 % Cream (Experimental): Participants received ruxolitinib 1.5% cream, applied topically to the affected area as defined in the protocol.
  Interventions: Drug: Ruxolitinib Cream
- Vehicle Cream (Placebo Comparator): Participants received vehicle cream, applied topically to the affected area as defined by the protocol.
  Interventions: Drug: Vehicle Cream

INTERVENTIONS:
Drug: Ruxolitinib Cream — Ruxolitinib cream applied topically to the affected area as a thin film twice daily.
  Arms: Ruxolitinib 1.5 % Cream
Drug: Vehicle Cream — Matching vehicle cream applied topically to the affected area as a thin film twice daily.
  Arms: Vehicle Cream

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ruxolitinib cream in participants with hidradenitis suppurativa.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HS for at least 6 months prior to screening visit.
* Mild to moderate HS (Hurley I or II) with the following at both screening and baseline visits:

  * A total AN count of at least 4, with no draining tunnels AND
  * Affecting at least 2 distinct anatomical areas
* Agreement to NOT use topical and systemic antibiotics for treatment of HS during the vehicle-controlled period.
* Agreement to NOT use topical antiseptics, including washes and leave-on products on the areas affected by HS lesions during the vehicle-controlled period and Weeks 16 to 20 of the extension period.
* Further inclusion criteria apply.

Exclusion Criteria:

* Body surface areas to be treated exceed 20% BSA at screening or baseline
* Presence of draining tunnels at screening or baseline.
* Medical history including current or history of certain infections, cancer, lymphoproliferative disorders and other medical conditions at the discretion of the investigator.
* Laboratory values outside of the protocol-defined criteria.
* Pregnant or lactating participants, or those considering pregnancy during the period of their study participation.
* Further exclusion criteria apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2026-10-09 (Estimated); Study Completion 2027-07-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who achieve Hidradenitis Suppurativa (HS) Clinical Response 75 (HiSCR75) from baseline | Week 16
  HiSCR75 is defined as at least a 75% reduction from baseline in the total abscess and/or inflammatory nodule (AN) count with no increase from baseline in abscess or draining tunnel count.

SECONDARY OUTCOMES:
Proportion of participants with ≥ 1 flare | Up to 16 weeks
  Defined as ≥ 25% increase in AN count with a minimum increase in total AN count of 2 relative to baseline.
Proportion of participants who achieve Skin Pain Numeric Rating Scale (NRS)30 among participants with baseline Skin Pain NRS score ≥ 3 | Week 16
  Participants with a Skin Pain score of at least 3 at baseline and who achieve Skin Pain NRS30, defined as at least a 30% reduction and at least 1-unit reduction from baseline in the Skin Pain NRS.
Treatment-IR Population: Proportion of participants who achieve Hidradenitis Suppurativa Clinical Response 75 (HiSCR75) from baseline | Week 16
  Treatment IR-Population defined as participants who had an inadequate response, intolerance, or contraindication to prior topical or systemic medications for HS. HiSCR75 is defined as at least a 75% reduction from baseline in the total AN count with no increase from baseline in abscess or draining tunnel count.
Treatment-IR Population: Proportion of participants with ≥ 1 HS flare | Up to 16 weeks
  Defined as ≥ 25% increase in total AN count with a minimum increase in AN count of 2 relative to baseline.
Treatment-IR Population: Proportion of participants who achieve Skin Pain Numeric Rating Scale (NRS)30 at Week 12 among participants with baseline Skin Pain NRS score ≥ 3 | Week 16
  Participants with a Skin Pain score of at least 3 at baseline and who achieve Skin Pain NRS30, defined as at least a 30% reduction and at least 1-unit reduction from baseline in the Skin Pain NRS.
Proportion of participants who achieve HiSCR50/75/90/100 at each postbaseline visit | Up to 16 weeks
  Defined as ≥ 50%/75%/90%/100% reduction from baseline in total AN count with no increase from baseline in abscess or draining tunnel count.
Extension Period: Proportion of participants with ≥ 1 HS flare | From Week 16 through Week 52
  Defined as ≥ 25% increase in total AN count with a minimum increase in AN count of 2 relative to baseline.
Proportion of participants who achieve abscess and/or inflammatory nodule (AN)75 at each postbaseline visit | Up to 52 weeks
  Defined as ≥ 75% reduction from baseline in total AN count.
Mean change from baseline in total AN count at each postbaseline visit | Up to 52 weeks
  Defined as mean change in total AN count.
Percentage change from baseline in total AN count at each postbaseline visit | Up to 52 weeks
  Defined as percent change from baseline in total AN count.
Mean change from baseline in abscess count at each postbaseline visit | Up to 52 weeks
  Defined as mean change of abscess(es) count relative to baseline.
Percentage change from baseline in abscess count at each postbaseline visit | Up to 52 weeks
  Percent Change from baseline in number of abscess(es).
Mean change from baseline in inflammatory nodule count at each postbaseline visit | Up to 52 weeks
  Defined as mean change of inflammatory nodule count relative to baseline.
Percentage change from baseline in inflammatory nodule count at each postbaseline visit | Up to 52 weeks
  Defined as percent change from baseline in number of inflammatory nodule(s).
Proportion of participants with presence of draining tunnels at each postbaseline visit | Up to 52 weeks
  Participants with presence of draining tunnels.
Proportion of participants who achieve Skin Pain Numeric Rating Scale (NRS)30 among participants with baseline Skin Pain NRS score ≥ 3 at each postbaseline visit | Up to 52 weeks
  Participants with a Skin Pain score of at least 3 at baseline and who achieve Skin Pain NRS30, defined as at least a 30% reduction and at least 1-unit reduction from baseline in the Skin Pain NRS.
Proportion of participants who achieve Itch Numeric Rating Scale (NRS)30 among participants with baseline Itch NRS score ≥ 3 at each postbaseline visit | Up to 52 weeks
  Participants with a Itch score of at least 3 at baseline and who achieve Itch NRS30, defined as at least a 30% reduction and at least 1-unit reduction from baseline in the Itch NRS.
Proportion of participants who achieve Patient Global Impression of Change (PGIC) at each postbaseline visit | Up to 52 weeks
  The PGIC is based on a 7-point scale and the participant will rate each question from the start of treatment as 1-very much improved, 2-much improved, 3-minimally improved, 4-no change, 5-minimally worse, 6-much worse, and 7-very much worse.
Proportion of participants who achieve PGIC score 1 or 2 at each postbaseline visit | Up to 52 weeks
  The PGIC is based on a 7-point scale and the participant will rate each question from the start of treatment as 1-very much improved, 2-much improved, 3-minimally improved, 4-no change, 5-minimally worse, 6-much worse, and 7-very much worse.
Patient Global Impression of Severity (PGIS) score at each postbaseline visit | Up to 52 weeks
  The PGIS is a single-item, self-reporting measure in which the participant rates the severity of their overall status over the past week based on a 5-point scale: (1) none, (2) mild, (3) moderate, (4) severe, and (5) very severe.
Change from baseline in PGIS Score at each postbaseline visit | Up to 52 weeks
  The PGIS is a single-item, self-reporting measure in which the participant rates the severity of their overall status over the past week based on 5-point scale: (1) none, (2) mild, (3) moderate, (4) severe, and (5) very severe.
Proportion of participants who achieve status of Dermatology Life Quality Index (DLQ1)4 at each postbaseline visit | Up to 52 weeks
  Defined as a ≥ 4-point reduction in DLQI score relative to baseline. The DLQI is a simple, 10-question, validated questionnaire to measure how much a skin problem has affected an adult participant over the previous 7 days, across symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment.
Proportion of participants who achieve status of Children's Dermatology Life Quality Index (CDLQ1)6 at each postbaseline visit | Up to 52 weeks
  Defined as a ≥ 6-point reduction in CDLQI score relative to baseline. The CDLQI is a 10-question, validated questionnaire to measure the impact of skin disease on the lives of children over the previous 7 days.
Change from baseline in Hidradenitis Suppurativa Quality of Life (HiSQoL) score at each postbaseline visit | Up to 52 weeks
  The HiSQoL is a 17-item, HS-specific, health-related, quality-of-life instrument with a 7-day recall period used to assess HS symptoms and the impact of HS problems on quality of life.
Percent change from baseline in Hidradenitis Suppurativa Quality of Life (HiSQoL) score at each postbaseline visit | Up to 52 weeks
  The HiSQoL is a 17-item, HS-specific, health-related, quality-of-life instrument with a 7-day recall period used to assess HS symptoms and the impact of HS problems on quality of life.
Change from baseline in Hidradenitis Suppurativa Quality of Life - Adolescent (HiSQoL-AA) at each postbaseline visit | Up to 52 weeks
  The HiSQoL-AA is a 15-item instrument with a 7-day recall period used to assess HS symptoms and experiences of HS in adolescent.
Percent change from baseline in Hidradenitis Suppurativa Quality of Life - Adolescent (HiSQoL-AA) at each postbaseline visit | Up to 52 weeks
  he HiSQoL-AA is a 15-item instrument with a 7-day recall period used to assess HS symptoms and experiences of HS in adolescent.
Change from baseline in EuroQol 5-dimension 5-level scale (EQ-5D-5L) score at each postbaseline visit | Up to 52 weeks
  The EQ-5D-5L questionnaire is a standardized, validated instrument for use as a measure of health outcome.
Treatment-IR Population: Change from baseline in total abscess count at each postbaseline visit | Up to 52 weeks
  Defined as change from baseline in total abscess count.
Treatment-IR Population: Percent change from baseline in total abscess count at each postbaseline visit | Up to 52 weeks
  Percent Change from baseline in total abscess count.
Treatment-IR Population: Change from baseline in total inflammatory nodule count at each postbaseline visit | Up to 52 weeks
  Defined as change from baseline in total number of inflammatory nodule(s).
Treatment-IR Population: Percent change from baseline in total inflammatory nodule count at each postbaseline visit | Up to 52 weeks
  Defined as percent change from baseline in number of inflammatory nodule(s).
Treatment-IR Population: Proportion of participants with presence of draining tunnels at each postbaseline visit | Up to 52 weeks
  Participants with presence of draining tunnels.
Number of Treatment Emergent Adverse Events (TEAEs) | Up to 56 weeks
  A TEAE or treatment emergent SAE is any AE or SAE either reported for first time or worsening of a pre-existing event after first application of study cream.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Study Monitor, Study Director — Incyte Corporation
Locations (106):
- United States (60):
  - Investigative Site US020, Phoenix, Arizona
  - Investigative Site US033, Scottsdale, Arizona
  - Investigative Site US054, Tempe, Arizona
  - Investigative Site US002, Fayetteville, Arkansas
  - Investigative Site US055, Brea, California
  - Investigative Site US004, Laguna Niguel, California
  - Investigative Site US007, Los Angeles, California
  - Investigative Site US013, San Diego, California
  - Investigative Site US060, San Diego, California
  - Investigative Site US038, San Diego, California
  - Investigative Site US059, Aurora, Colorado
  - Investigative Site US045, Boynton Beach, Florida
  - Investigative Site US028, Fort Myers, Florida
  - Investigative Site US016, Miami, Florida
  - Investigative Site US027, Sanford, Florida
  - Investigative Site US057, Sweetwater, Florida
  - Investigative Site US029, Tampa, Florida
  - Investigative Site US061, Atlanta, Georgia
  - Investigative Site US053, Atlanta, Georgia
  - Investigative Site US019, Marietta, Georgia
  - Investigative Site US026, Chicago, Illinois
  - Investigative Site US049, Clarksville, Indiana
  - Investigative Site US052, West Lafayette, Indiana
  - Investigative Site US001, Bowling Green, Kentucky
  - Investigative Site US022, Louisville, Kentucky
  - Investigative Site US050, Baton Rouge, Louisiana
  - Investigative Site US046, Glenn Dale, Maryland
  - Investigative Site US003, Boston, Massachusetts
  - Investigative Site US030, Boston, Massachusetts
  - Investigative Site US010, Quincy, Massachusetts
  - Investigative Site US051, Detroit, Michigan
  - Investigative Site US006, Minneapolis, Minnesota
  - Investigative Site US021, New Brighton, Minnesota
  - Investigative Site US036, Saint Joseph, Missouri
  - Investigative Site US034, New City, New York
  - Investigative Site US018, New York, New York
  - Investigative Site US017, New York, New York
  - Investigative Site US023, Rochester, New York
  - Investigative Site US014, Chapel Hill, North Carolina
  - Investigative Site US025, Fargo, North Dakota
  - Investigative Site US015, Bexley, Ohio
  - Investigative Site US044, Cincinnati, Ohio
  - Investigative Site US008, Columbus, Ohio
  - Investigative Site US031, Mason, Ohio
  - Investigative Site US048, Oklahoma City, Oklahoma
  - Investigative Site US043, Danville, Pennsylvania
  - Investigative Site US056, Philadelphia, Pennsylvania
  - Investigative Site US024, Charleston, South Carolina
  - Investigative Site US041, Myrtle Beach, South Carolina
  - Investigative Site US005, Murfreesboro, Tennessee
  - Investigative Site US047, Nashville, Tennessee
  - Investigative Site US062, Dallas, Texas
  - Investigative Site US035, El Paso, Texas
  - Investigative Site US032, Frisco, Texas
  - Investigative Site US012, Plano, Texas
  - Investigative Site US011, San Antonio, Texas
  - Investigative Site US040, Layton, Utah
  - Investigative Site US037, Murray, Utah
  - Investigative Site US039, Ogden, Utah
  - Investigative Site US058, Seattle, Washington
- Bulgaria (2):
  - Investigative Site BG002, Sofia
  - Investigative Site BG003, Sofia
- Canada (9):
  - Investigative Site CA004, Calgary, Alberta
  - Investigative Site CA003, Calgary, Alberta
  - Investigative Site CA009, Ottawa, Ontario
  - Investigative Site CA002, Peterborough, Ontario
  - Investigative Site CA001, Richmond Hill, Ontario
  - Investigative Site CA007, Toronto, Ontario
  - Investigative Site CA005, Toronto, Ontario
  - Investigative Site CA006, Waterloo, Ontario
  - Investigative Site CA008, Sherbrooke, Quebec
- France (5):
  - Investigative Site FR002, Bordeaux
  - Investigative Site FR005, Brest
  - Investigative Site FR004, Nantes
  - Investigative Site FR003, Nice
  - Investigative Site FR001, Paris
- Germany (8):
  - Investigative Site DE006, Berlin
  - Investigative Site DE005, Berlin
  - Investigative Site DE002, Bochum
  - Investigative Site DE004, Darmstadt
  - Investigative Site DE001, Dresden
  - Investigative Site DE003, Erlangen
  - Investigative Site DE007, Hamburg
  - Investigative Site DE008, Lübeck
- Italy (9):
  - Investigative Site IT001, Catania
  - Investigative Site IT005, Cona
  - Investigative Site IT009, Florence
  - Investigative Site IT003, Milan
  - Investigative Site IT007, Naples
  - Investigative Site IT006, Roma
  - Investigative Site IT004, Roma
  - Investigative Site IT002, Rozzano
  - Investigative Site IT008, Torino
- Poland (4):
  - Investigative Site PL002, Lodz
  - Investigative Site PL003, Torun
  - Investigative Site PL001, Warsaw
  - Investigative Site PL004, Wroclaw
- Spain (5):
  - Investigative Site ES004, Alicante
  - Investigative Site ES005, Badalona
  - Investigative Site ES003, Barcelona
  - Investigative Site ES001, Madrid
  - Investigative Site ES002, Madrid
- United Kingdom (4):
  - Investigative Site GB001, Cardiff
  - Investigative Site GB004, Harrogate
  - Investigative Site GB002, Ipswich
  - Investigative Site GB006, London

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: Study to Evaluate the Efficacy and Safety of Ruxolitinib Cream in Participants With Hidradenitis Suppurativa (TRuE-HS1) — https://incyteclinicaltrials.com/studies/incb018424-324